CLINICAL TRIAL: NCT02505802
Title: Phase III Study of Botulinum Toxin A Injection for Lower Limbs Spasticity in Subacute Stroke Adults
Brief Title: The Effectiveness of Early Botulinum Toxin A Injection for Lower Limbs Spasticity in Subacute Stroke Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, TAO WU, MD, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013KYB163
Record Dates: First submitted 2015-07-17; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Stroke; Muscle Spasticity
Keywords: Stroke; Botulinum Toxins; Muscle Spasticity; Gait
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BoNT-A treatment group (Experimental): In BoNT-A treatment group patients received 200 units BoNT-A injection in the triceps surae (150iu) and tibial muscle posterior (50iu). Both groups received comprehensive rehabilitation for 8 weeks.
  Interventions: Drug: BoNT-A injection
- Control group (No Intervention): No special treatment was performed in the control group. Both groups received comprehensive rehabilitation for 8 weeks.

INTERVENTIONS:
Drug: BoNT-A injection — In BoNT-A treatment group patients received 200 units BoNT-A injection in the triceps surae (150iu) and tibial muscle posterior (50iu).
  Other Names: Botulinum toxin A
  Arms: BoNT-A treatment group

SUMMARY:
Botulinum toxin A (BoNT-A) injections are widely used to treat spasticity after stroke. Although this treatment is effective on muscle tone improvement, its effect on gait and ability of daily living on early stage of stroke adults remains uncertain.The purpose of this study is to determine whether an early calf muscle injection of low dose BoNT-A in severely affected patients within 6 weeks after stroke could help to hold back disabling muscle spasticity and improve walking dysfunction.

DETAILED DESCRIPTION:
The high prevalence of stroke is a global problem causing well-known long-term disabilities. Post-stroke lower-extremity spasticity may cause severe functional limitations and pain. Spasticity is a phenomenon defined as disordered sensory-motor control, resulting from upper motor neuron (UMN) lesion, presenting as intermittent or sustained involuntary activation of muscles . Spasticity may interfere with motor function, and is a common reason for clinical interventions such as by physiotherapy, use of orthoses or other technical devices or drugs. Botulinum toxin A (BoNT-A) is a potent neurotoxin that is produced by the bacterium clostridium botulinum. BoNT-A, by blocking acetylcholine release at neuromuscular junctions, accounts for its therapeutic action to relieve dystonia, spasticity, and related disorders.

Unfortunately, intramuscular injections of botulinum often carried out when the patients have obvious spasticity . It is normally given until the clinical signs of an elevated muscle tone have become established; therefore it is usually given at least three months after stroke , . It will impede the rehabilitation of the patients. Accordingly, the present study asked whether an early calf muscle injection of low dose BoNT-A in severely affected patients within 6 weeks after stroke could help to hold back disabling muscle spasticity and improve walking dysfunction along 24 weeks fellow up trail.

This is a randomized, open-label, controlled trial along 24-weeks trails. Referred sample of adult subacute stroke patients (within 6 weeks since stroke, n=30) with mild spasticity of calf muscle will be included. Patients were randomly allocated to BoNT-A treatment group (15 patients) and control group (15 patients). In BoNT-A treatment group patients received 200 units BoNT-A injection in the triceps surae (150iu) and tibial muscle posterior (50iu). No special treatment was performed in the control group. Both groups received comprehensive rehabilitation for 8 weeks. Lower limbs Fugl-Meyer (FM) score, calf muscle modified Ashworth scale assess (MAS), gastrocnemius surface electromyography (sEMG) evaluation and modified Barthel index (MBI) were assessed before and 8, 12, 24 weeks after treatment. Gait analysis (step length，cadence，speed), 6-min walking distance were assessed 8, 12, 24 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Were over the age of 18 and less than 80 years and had a stroke within 6 weeks.
2. Had slight spasticity of the triceps surae as defined by a score of 1-1+ on the Modified Ashworth Scale (MAS) or ankle clonus (+).
3. Had sufficient cognitive and communication ability as defined by MMSE (mini-mental state examination)>25.
4. Couldn't dorsiflex ankle and their LEMI (Lower Extremity Motor Index) < 10.
5. Were not receiving concurrent aminoglycoside antibiotics and oral anti-spasticity medication

Exclusion Criteria:

1. Known allergy or sensitivity to study medication or its components.
2. Infection or dermatological condition at the injection sites.
3. Any medical condition that may put the subject at increased risk with exposure , including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might have interfered with neuromuscular function.
4. QTc criteria: QTc ≥ 450 millisecond (msec) or≥480msec for subjects with Bundle Branch Block-values based on either single electrocardiogram (ECG) values or triplicate ECG averaged QTc values obtained over a brief recording period
5. Liver function tests: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥2xULN; alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
6. Concurrent use of aminoglycoside antibiotics or other agents that might interfere with neuromuscular function.
7. Patients with severe cognitive impairment or neurological diseases affecting the implementation or evaluation of the test, and drug-dependent patients.
8. Presence of clinically unstable severe cardiovascular, renal or respiratory disease
9. Researchers believe there are other factors unfit to participate in this study of patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Calf muscle modified Ashworth scale assess (MAS) | The outcome will be undertaken at weeks 0 (baseline), 8, 12 and 24 weeks later

SECONDARY OUTCOMES:
Lower limbs Fugl-Meyer (FM) score | The outcome will be undertaken at weeks 0 (baseline), 8, 12 and 24 weeks later
Average integrated sEMG levels of gastrocnemius | The outcome will be undertaken at weeks 0 (baseline), 8, 12 and 24 weeks later
  Average integrated surface electromyography (sEMG) levels of gastrocnemius during the slow passive dorsiflexion of the ankle.
6-min walking distance | The outcome will be were assessed 8, 12, 24 weeks after injection.
Gait analysis (step length，cadence，speed). | The outcome will be undertaken at weeks 0 (baseline), 8, 12 and 24 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: TAO WU, MD, Study Director — Sir Run Run Shaw Hospital, College of Medicine, Zhejiang University
Locations (1):
- Sir Run Run Shaw Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Lundstrom E, Terent A, Borg J. Prevalence of disabling spasticity 1 year after first-ever stroke. Eur J Neurol. 2008 Jun;15(6):533-9. doi: 10.1111/j.1468-1331.2008.02114.x. Epub 2008 Mar 18. PMID 18355307
- [Result] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Result] McIntyre A, Lee T, Janzen S, Mays R, Mehta S, Teasell R. Systematic review of the effectiveness of pharmacological interventions in the treatment of spasticity of the hemiparetic lower extremity more than six months post stroke. Top Stroke Rehabil. 2012 Nov-Dec;19(6):479-90. doi: 10.1310/tsr1906-479. PMID 23192713
- [Result] Kaji R, Osako Y, Suyama K, Maeda T, Uechi Y, Iwasaki M; GSK1358820 Spasticity Study Group. Botulinum toxin type A in post-stroke lower limb spasticity: a multicenter, double-blind, placebo-controlled trial. J Neurol. 2010 Aug;257(8):1330-7. doi: 10.1007/s00415-010-5526-3. Epub 2010 Apr 1. PMID 20358216
- [Result] Cosgrove AP, Graham HK. Botulinum toxin A prevents the development of contractures in the hereditary spastic mouse. Dev Med Child Neurol. 1994 May;36(5):379-85. doi: 10.1111/j.1469-8749.1994.tb11863.x. PMID 8168656
- [Result] Santamato A, Micello MF, Panza F, Fortunato F, Pilotto A, Giustini A, Testa A, Fiore P, Ranieri M, Spidalieri R. Safety and efficacy of incobotulinum toxin type A (NT 201-Xeomin) for the treatment of post-stroke lower limb spasticity: a prospective open-label study. Eur J Phys Rehabil Med. 2013 Aug;49(4):483-9. Epub 2013 Mar 13. PMID 23480980